CLINICAL TRIAL: NCT00099346
Title: A Phase I/IIa Study Evaluating the Safety/Tolerability, Pharmacokinetics, and Efficacy of MK0457 Administered as a 5-Day Continuous Infusion in Patients With Advanced Colorectal Cancer and Other Solid Tumors
Brief Title: MK0457 (an Aurora Kinase Inhibitor) Study in Patients With Advanced Colorectal Cancer and Other Advanced Solid Tumors (0457-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0457-001; MK0457-001; 2004_095
Record Dates: First submitted 2004-12-10; First posted 2004-12-13 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Cancer; Advanced Solid Tumors
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tozasertib

INTERVENTIONS:
Drug: MK0457, VX-680 (Aurora Kinase Inhibitor)

SUMMARY:
Study with an investigational drug in patients with recurrent or non-responsive colorectal cancer or other advanced solid tumors.

This is an early phase trial and some specific protocol information is proprietary and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* In Part I, patients who are at least 18 years of age with advanced solid tumors and colorectal cancer will be eligible for the first part of this study. Patient must have recovered from and be at least 3 weeks from previous cancer treatment.
* In Part II, only patients with colorectal cancer will be eligible to participate. The patients may have received up to 3 prior treatments for their colorectal cancer. Patients must have recovered from and be at least 3 weeks from previous therapy.

Exclusion Criteria:

* Patients who have had treatment with any investigational drug within the past 30 days.
* Patients who have certain types of blood cancers such as leukemia or lymphoma.
* Patients who have uncontrolled congestive heart failure (CHF), chest pain, or heart attack within the past 3 months.
* Patient is pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC